CLINICAL TRIAL: NCT07033494
Title: A Phase 2 Randomized, Placebo-Controlled, Double-Blind, Parallel-Group Study to Evaluate the Efficacy and Safety of MK-2214 in Participants With Early Alzheimer's Disease
Brief Title: A Clinical Study of MK-2214 in People With Early Alzheimer's Disease (MK-2214-004)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2214-004; MK-2214-004 (Other: MSD); 2024-519190-19-00 (Registry Identifier: EU CT); U1111-1314-8296 (Registry Identifier: UTN); jRCT2031250299 (Registry Identifier: Japan Registry of Clinical Trial (jRCT))
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Early Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-2214 (Experimental): Participants will receive MK-2214 via intravenous (IV) infusion every 4 weeks (q4w) during the study.
  Interventions: Biological: MK-2214
- Placebo (Placebo Comparator): Participants will receive a placebo via IV infusion q4w during the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: MK-2214 — IV infusion
  Arms: MK-2214
Drug: Placebo — IV infusion
  Arms: Placebo

SUMMARY:
Researchers want to know if the study treatment called MK-2214 works to slow certain changes in the brains of people with Alzheimer's disease (AD). AD is a type of dementia that can cause loss of memory, communication (such as speech), and decision-making skills. It can limit a person's ability to do daily tasks. MK-2214 is a study treatment designed to slow down AD.

The goals of the study are to learn:

* If MK-2214 slows the spread of tau in the brain compared to placebo. Tau is a protein that accumulates in AD & damages brain cells. A placebo looks like the study treatment but has no study treatment in it. Using a placebo helps researchers better understand the effects of a study treatment.
* About the safety of MK-2214 and if people tolerate it

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has mild cognitive impairment (MCI) or mild dementia due to Alzheimer's Disease (AD)
* Has a designated study partner who can fulfill the requirements of this study
* If on an approved AD therapy for symptomatic AD, the dosing regimen must have been stable for 3 months prior to screening

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a known history of stroke or cerebrovascular disease
* Has diagnosis of a clinically relevant central nervous system disease other than AD or other condition that negatively impacts cognition or cognitive status chronically
* Has structural brain disease
* Has a history of seizures or epilepsy within 5 years before screening
* Has any other major central nervous system trauma, or infections that affect brain function
* Has major medical illness or unstable medical condition within 3 months before screening
* Has a severe, acute, or chronic medical or psychiatric condition or laboratory abnormality
* Has any immunological disease, which is not adequately controlled, or which requires treatment with biologics and/or immunosuppressants during the study
* Has a bleeding disorder that is not under adequate control
* Has a history of malignancy occurring within 5 years of screening
* Has a risk factor for corrected QT interval (QTc) prolongation
* Has liver disease
* Is unwilling or unable to undergo computed tomography (CT), positron emission tomography (PET), or magnetic resonance imaging (MRI) scan
* Resides in a nursing home or assisted care facility with need for direct continuous medical care and nursing supervision

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Tau PET Standardized Uptake Value Ratio (SUVr) | Baseline, up to approximately 23 months
  Participants will have tau PET imaging to assess tau pathology. Tau is a protein that accumulates in AD & damages brain cells. SUVr is SUV in the region of interest divided by SUV in a reference region (cerebellum). The change from baseline in tau PET SUVr will be reported.
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 26 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience one or more AEs will be reported.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 23 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study intervention due to an AE will be reported.

SECONDARY OUTCOMES:
Change from Baseline in the Clinical Dementia Rating-Sum of Boxes (CDR-SB) Total Score | Baseline, up to approximately 23 months
  The CDR-SB is used for cognitive assessment in people with AD. The CDR is a clinical scale that describes 5 degrees of impairment in performance on each of 6 categories of function including memory, orientation, judgment and problem solving, community affairs, home and hobbies, and personal care. The ratings of degree of impairment obtained on each of the 6 categories of function are synthesized into 1 global rating of dementia CDR score ranging from 0 (normal) to 3 (severe). A total score is calculated as the sum of the category scores, with a range of 0 (normal) to 18 (severe). Higher scores indicate more impairment. The change from baseline in CDR-SB total score will be reported.
Change from Baseline in the Composite Tau PET SUVr in Braak Region III and IV | Baseline, up to approximately 23 months
  Participants will have tau PET imaging to assess tau pathology. Tau is a protein that accumulates in AD & damages brain cells. SUVr is SUV in the region of interest, divided by SUV in a reference region (cerebellum). Braak staging ranges from Braak I to VI. Description for Braak III includes amygdala, parahippocampal gyrus, fusiform gyrus, & lingual gyrus, and Braak IV includes insula, inferior temporal, lateral temporal, posterior cingulate, & inferior parietal. The composite tau PET SUVr is a weighted average of tau PET SUVr values obtained from multiple brain regions, with weights being the percentage volume of each region within the composite. The change from baseline in composite tau PET SUVr in Braak regions III and IV will be reported.
Change from Baseline in the Composite Tau PET SUVr | Baseline, up to approximately 23 months
  Participants will have tau PET imaging to assess tau pathology. Tau is a protein that accumulates in AD & damages brain cells. SUVr is SUV in the region of interest, divided by SUV in a reference region (cerebellum). The composite tau PET SUVr is a weighted average of tau PET SUVr values obtained from multiple brain regions, with weights being the percentage volume of each region within the composite. The change from baseline in composite tau PET SUVr will be reported.
Change from Baseline in the Composite Tau PET SUVr in Braak Region I to VI | Baseline, up to approximately 23 months
  Participants will have tau PET imaging to assess tau (protein that accumulates in AD & damages brain cells) pathology. SUVr is SUV in the region of interest, divided by SUV in a reference region (cerebellum). Braak staging ranges from I-VI (Braak I (transentorhinal); II (entorhinal & hippocampus); III (amygdala, parahippocampal gyrus, fusiform gyrus, & lingual gyrus); IV (insula, inferior temporal, lateral temporal, posterior cingulate, & inferior parietal); V (orbitofrontal, superior temporal, inferior frontal, cuneus, anterior cingulate, supramarginal gyrus, lateral occipital, precuneus, superior parietal, superior frontal, & rostro medial frontal); VI (paracentral, postcentral, precentral, & pericalcarine)). Composite tau PET SUVr is weighted average of tau PET SUVr values from multiple brain regions, with weights being percentage volume of each region. The change from baseline in composite tau PET SUVr in Braak region I to IV will be reported.
Change from Baseline in the Alzheimer's Disease Assessment Scale-Cognitive Subscale13 (ADAS-Cog13) Total Score | Baseline, up to approximately 23 months
  The ADAS-Cog13 is a structured scale that evaluates memory (word recall, delayed word recall, and word recognition), reasoning (following commands), language (naming, comprehension), orientation, ideational praxis (placing letter in envelope) and constructional praxis (copying geometric designs). In addition, ratings of spoken language, language comprehension, word finding difficulty, ability to remember test instructions, and number cancellation will be obtained. Per protocol, score range will be from 0 (no impairment) to 85 (maximum impairment) points. Higher scores indicate more impairment. The change from baseline in ADAS-Cog13 total score will be reported.
Change from Baseline in the Alzheimer's Disease Cooperative Study Activities of Daily Living for Mild Cognitive Impairment (ADCS-ADL-MCI) Total Score | Baseline, up to approximately 23 months
  ADCS-ADL-MCI evaluates the ability of individuals to perform various daily activities including basic activities of daily living (BADL; personal care tasks like bathing, dressing and eating) and instrumental activities of daily living (IADL; complex tasks such as managing finances, preparing meals, using telephone) administered through caregiver or family member to access severity of cognitive decline in the past 4 weeks. Each item is scored on a scale of 0 (unable to do) to 2 (independent). The total score is calculated by summing scores of all items and ranges from 0 (poor functioning) to 68 (better functioning). Higher scores indicate better functional ability. The change from baseline in ADCS-ADL-MCI total score will be reported.
Change from Baseline in Modified Integrated Alzheimer's Disease Rating Scale (iADRS) Total Score | Baseline, up to approximately 23 months
  The modified iADRS is a composite tool to measure cognition and function. The modified iADRS is a linear combination of total scores from the ADAS-Cog and the ADCS-ADL-MCI. The modified iADRS composite score is calculated by subtracting the ADAS-Cog13 score from 85 and then adding the ADCS-ADL-MCI score. Composite score ranges from 0 (maximum impairment) to 144 (greater independent, healthy functioning and cognition). Lower scores indicate more impairment. The change from baseline in modified iADRS total score will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (68):
- United States (35):
  - Inglewood Clinical ( Site 1062), Inglewood, California
  - Irvine Clinical Research ( Site 1041), Irvine, California
  - Healthy Brain Clinic ( Site 1005), Long Beach, California
  - Anderson Clinical Research ( Site 1024), Redlands, California
  - UCSF Memory and Aging Center ( Site 1031), San Francisco, California
  - Syrentis Clinical Research ( Site 1001), Santa Ana, California
  - Yale University, Alzheimer's Disease Research Unit ( Site 1059), New Haven, Connecticut
  - JEM Research Institute ( Site 1046), Atlantis, Florida
  - Neuropsychiatric Research Center of Southwest Florida ( Site 1003), Fort Myers, Florida
  - Indago Research & Health Center, Inc ( Site 1044), Hialeah, Florida
  - K2 Medical Research ( Site 1047), Maitland, Florida
  - ClinCloud LLC ( Site 1039), Melbourne, Florida
  - Aqualane Clinical Research ( Site 1035), Naples, Florida
  - Suncoast Clinical Research ( Site 1007), New Port Richey, Florida
  - Renstar Medical Research ( Site 1012), Ocala, Florida
  - Charter Research - Orlando ( Site 1051), Orlando, Florida
  - Axiom Brain Health ( Site 1029), Tampa, Florida
  - K2 Medical Research ( Site 1020), Tampa, Florida
  - Charter Research - Lady Lake ( Site 1019), The Villages, Florida
  - Conquest Research LLC ( Site 1053), Winter Park, Florida
  - CenExel iResearch, LLC ( Site 1015), Decatur, Georgia
  - Alexian Brothers Medical Center-Neurosciences ( Site 1017), Elk Grove Village, Illinois
  - Boston Center for Memory ( Site 1008), Newton, Massachusetts
  - Clinical Research Professionals ( Site 1004), Chesterfield, Missouri
  - The Cognitive and Research Center of New Jersey - Ridgewood ( Site 1064), Ridgewood, New Jersey
  - The Cognitive and Research Center of NJ ( Site 1057), Springfield, New Jersey
  - CenExel- AMRI ( Site 1018), Toms River, New Jersey
  - Alzheimer Disease Research Center (ADRC) ( Site 1000), Albany, New York
  - Mid Hudson Medical Research ( Site 1050), New Windsor, New York
  - Basil Clinical ( Site 1065), Queens, New York
  - Insight Clinical Trials ( Site 1011), Independence, Ohio
  - Neuro-Behavioral Clinical Research ( Site 1028), North Canton, Ohio
  - Flourish Research ( Site 1048), Plymouth Meeting, Pennsylvania
  - Gadolin Research ( Site 1032), Beaumont, Texas
  - Horizon Clinical Research Center - Houston ( Site 1026), Cypress, Texas
- Argentina (2):
  - Organizacion Medica de Investigacion ( Site 0401), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (FLENI) ( Site 0400), Caba
- Australia (3):
  - Southern Neurology ( Site 0306), Kogarah, New South Wales
  - KARA Institute for Neurological Diseases ( Site 0302), Macquarie Park, New South Wales
  - Austin Health ( Site 0300), Ivanhoe, Victoria
- Belgium (2):
  - UZ Leuven ( Site 3000), Leuven, Vlaams-Brabant
  - AZ Groeninge Campus Kennedylaan ( Site 3002), Kortrijk, West-Vlaanderen
- Japan (10):
  - National Center for Geriatrics and Gerontology ( Site 9002), Ōbu, Aichi-ken
  - Chibaken Saiseikai Narashino Hospital ( Site 9000), Narashino, Chiba
  - Association of Healthcare Corporation Koukankai Koukan Clinic ( Site 9016), Kawasaki, Kanagawa
  - Mie University Hospital ( Site 9011), Tsu, Mie-ken
  - Katayama Medical Clinic ( Site 9005), Kurashiki, Okayama-ken
  - National Hospital Organization Hizen Psychiatric Medical Center ( Site 9004), Kanzaki-gun, Saga-ken
  - Tokyo Medical University Hospital ( Site 9003), Shinjuku, Tokyo
  - Inage Neurology and Memory Clinic ( Site 9001), Chiba
  - Kyushu University Hospital ( Site 9010), Fukuoka
  - Okayama City General Medical Center Okayama City Hospital ( Site 9008), Okayama
- Netherlands (3):
  - Brain Research Center Den Bosch B.V. ( Site 5001), 's-Hertogenbosch, North Brabant
  - Brain Research Center. ( Site 5000), Amsterdam, North Holland
  - Brain Research Center Zwolle ( Site 5002), Zwolle, Overijssel
- South Korea (3):
  - Hanyang University Hospital ( Site 0200), Seoul
  - Samsung Medical Center ( Site 0202), Seoul
  - Ewha Womans University Seoul Hospital ( Site 0201), Seoul
- Spain (4):
  - Hospital Universitari Mutua Terrassa ( Site 6004), Terrassa, Barcelona
  - Fundació ACE ( Site 6003), Barcelona, Catalonia
  - Hospital del Mar ( Site 6001), Barcelona
  - Hospital Clinic i Provincial ( Site 6002), Barcelona
- United Kingdom (6):
  - Scottish Brain Sciences Aberdeen ( Site 8001), Aberdeen, Aberdeen City
  - Scottish Brain Sciences ( Site 8000), Edinburgh, Edinburgh, City of
  - Moorgreen Hospital ( Site 8004), Southampton, Hampshire
  - Warneford Hospital ( Site 8007), Oxford, Oxfordshire
  - Remind UK ( Site 8003), Bath, Somerset
  - Re:Cognition Health - Birmingham ( Site 8002), Birmingham

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com